CLINICAL TRIAL: NCT02096796
Title: Hand Strength Grip and Ergonomics of Driving as Risk Factors in the Etiology of Arm Pump in Motorcross Training
Brief Title: Arm Pump in Motorcross Training
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Prof. Dr. F. Staes, Professor, Universitaire Ziekenhuizen KU Leuven
Other Study IDs: S56412
Record Dates: First submitted 2014-03-21; First posted 2014-03-26 (Estimated); Last update posted 2015-09-17 (Estimated); Status verified 2015-09

CONDITIONS: Healthy Individuals; Patients With Arm Pump

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- persons without arm pump
- persons with arm pump

SUMMARY:
Arm Pump is a sport specific term drivers use to describe Acute or Chronic Compartment Syndrome of the forearm. Drivers experience pain in the forearms due to increased blood pressure in forearm muscle compartments. No strategies nor methods have been used to diminish the risk to suffer from arm pump within motor cross.

This project aims to look at ergonomics of driving and its relationship with the occurrence of arm pump.

The investigators will first investigate the experience of motor cross athletes with arm pump through motor cross federations in Belgium and The Netherlands (survey).

Two groups of athletes will be selected (20 persons within each group) who will be invited to the motor cross track to investigate their hand grip strength, motor driving position, muscle activity.

ELIGIBILITY:
Inclusion Criteria:

* recreational or competitive motor cycling athletes
* with or without arm pump problems
* signing informed consent
* participation with their own motor bike
* Regular training hours

Exclusion Criteria:

* Inactive for more than 2 weeks before participation
* Pathology at shoulder, elbow or wrist level (except for arm pump)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Recreational or competitive motor cycle athletes
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2014-04; Primary Completion 2014-12 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
motor ergonomics | March - June 2014 (3 months)
  2D video-recording will be used to observe motor sitting position

SECONDARY OUTCOMES:
hand grip strength | March - June 2014 (3 months)
  Use of hand grip dynamometer (Biometrics) to measure hand grip strength.

OTHER OUTCOMES:
muscle activity | March - June 2014 (3 months)
  Use of surface electromyography in order to record muscle activity of forearm and upper arm musculature

CONTACTS AND LOCATIONS:
Locations (1):
- Motor Cross Track, Lommel, Limbur, Belgium